CLINICAL TRIAL: NCT05402150
Title: Evaluation of an Online Intervention Targeting Depression and Low Reward Sensitivity - A Randomized Controlled Trial
Brief Title: An Online Intervention Targeting Depression and Low Reward Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ReSet your Mind
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Depression Mild; Depression Moderate
Keywords: reward sensitivity; reward processing; depression; randomized controlled trial; online intervention; behavioral activation; mindfulness; gratitude
MeSH Terms: conditions — Depression | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Behavioral Activation (Experimental): 14 days of daily excercises
  Interventions: Behavioral: Behavioral Activation
- Mindfulness and Gratitude (Experimental): 14 days of daily excercises
  Interventions: Behavioral: Mindulness and Gratitude
- Combination: Behavioral Activation and Mindfulness and Gratitude (Experimental): 14 days of daily excercises
  Interventions: Behavioral: Combination of Behavioral Activation and Mindfulness and Gratitude
- Waitlist control group (No Intervention): Will receive the intervention (combination) after two weeks of intervention time of the other groups.

INTERVENTIONS:
Behavioral: Behavioral Activation — * instruction to create a list of individual positive activities.
  * instruction to include daily positive activities and fill out a mood protocol, which covers the time period shortly before, during and after the activity.
  Arms: Behavioral Activation
Behavioral: Mindulness and Gratitude — * instruction to fill out a mindfulness diary: reflection of daily pleasant situation, instructing the participants to revisit the impressions of their 5 senses during this situation, in addition they should specify how long they have actually dealt with these pleasant impressions of the situation they reflected upon
  * instruction to do a gratitude exercise and name one or more things they are generally grateful for each day.
  Arms: Mindfulness and Gratitude
Behavioral: Combination of Behavioral Activation and Mindfulness and Gratitude — This group will do a combination of the two intervention types.
  Arms: Combination: Behavioral Activation and Mindfulness and Gratitude

SUMMARY:
This study aims to evaluate and compare the effectiveness of different online interventions targeting reward sensitivity and depressive symptoms. We hypothesize that behavioral activation, a mindfulness and gratitude intervention, as well as a combination of both, will significantly reduce depressive symptoms and increase reward sensitivity, compared to the waitlist group. In addition, we assume that behavioral activation will have an increased effect on reward sensitivity compared to the mindfulness and gratitude intervention.

The investigators will further investigate factors influencing treatment success in another paper based on data of this study (see secondary and other pre-specified outcome measures).

DETAILED DESCRIPTION:
Depression is characterized by low reward sensitivity, which is a potential maintaining factor of depressive symptoms. This is why treatment for depression should include evidence-based interventions that target reward insensitivity. Up until now, there is a lack of research that studies reward sensitivity as main outcome measure or focus of interventions, especially in the online format. However, it is crucial to identify psychological interventions that are most effective in treating low reward sensitivity. Previous studies showed that behavioral activation can be a powerful intervention to increase the availability of rewards in everyday life. In addition, mindfulness-based interventions offer effective interventions with regards to low reward sensitivity since mindfulness refocusses attention on the present moment.

This study aims to evaluate the effectiveness of different online interventions compared to a waitlist control condition in a randomized controlled trial. The sample will include participants with mild to moderate depressive symptoms, who have been preselected for their low trait reward responsiveness. Inclusion and exclusion criteria will be confirmed via a preliminary online survey and a telephone screening, which will be administered by a trained psychologist. Suicidal participants or participants who suffer from severe depression will be excluded. Those will be informed about possibilities to get intensive professional help. Further exclusion criteria will be an ongoing psychotherapy, an antidepressant medication which has been taken for a shorter time period than four weeks, persons with a lifetime diagnosis of bipolar disorder (I and II), psychotic disorders or a substance use disorder.

Participants will be randomly assigned into four groups. The randomization will be stratified according to their depression score (mild or moderate). The investigators aim to include 50 participants per group (N = 200 in total). The first group ("Behavioral Activation") will be instructed to include daily positive activities and fill out a mood protocol, which covers the time period shortly before, during and after the activity. The second group ("Mindfulness and Gratitude") will fill out a mindfulness diary and reflect upon daily pleasant situation via revisiting the impressions of their five senses during this situation. In addition, participants will specify how long they have dealt with the situation and will name something they are grateful for. The third group will do a combination of the two interventions. The fourth group will be the waitlist control condition and receive the intervention material of the third group after two weeks.

Participants will receive a pre-intervention online survey with questionnaires as a baseline measurement. This survey includes a psychoeducation video and an instruction video explaining the intervention rationale and the daily excercises. Participants will receive working sheets to protocol their daily exercises over a course of two weeks. In addition, participants are encouraged to report their results and possible problems with the implementation of the excercises in a short online survey. In addition, every day a different case study will be presented which deals with obstacles and shows strategies to solve problems. Furthermore, participants are able to contact the principal contact person of the study (Laura Potsch) via telephone to help with problems. After two weeks of daily interventions, participants will receive a post-questionnaire to measure treatment effects and will receive a follow up questionnaire after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Fluent in German
* Informed consent
* Depressive symptoms (PHQ-9 > 5)

Exclusion Criteria:

* suicidality, severe depression
* current or lifetime: substance use disorder, psychotic disorders, bipolar I or II
* current psychotherapy
* if antidepressant medication: has not been stable over the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms (Patient Health Questionnaire-9, PHQ-9) | baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 0 to 3 (0 = not at all; 1 = several days; 2 = more than a week; 3 = nearly every day).
  * PHQ-9 total score ranges from 0 to 27 (classification of scores: 5-9 mild depression; 10-14 as moderate depression; 15-19: moderately severe depression; 20 - 27 severe depression).
  * Consequently, a higher score means worse depressive symptoms.
Change in reward sensitivity (Positive Valence System Scale-21, PVSS-21) | baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 1 to 9 (1 = extremely untrue of me, 2 = very untrue of me, 3 = moderately untrue of me, 4 = slightly untrue of me, 5 = neutral, 6 = slightly true of me, 7 = moderately true of me, 8 = very true of me, 9 = extremely true of me).
  * PVSS-21 total score ranges from 21 to 189.
  * Consequently, a higher score means a higher reward responding.

SECONDARY OUTCOMES:
Somatization psychopathology (Patient Health Questionnaire-15, PHQ-15) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items in the PHQ-15 range from 0 to 2 (0 = not bothered at all, 1 = bothered a little, 2 = bothered a lot), two items (which are included in the PHQ-9 (question 2c and d) originally range from 0 to 3 (0 = not at all; 1 = several days; 2 = more than a week; 3 = nearly every day), here 2 and 3 are counted as 2.
  * PHQ-15 total score ranges from 0 to 30 (classification of scores: ≥5 mild level of somatization, ≥10 moderate level of somatization, ≥15 severe level of somatization).
  * Consequently, a higher score means a worse somatization.
Generalized anxiety disorder psychopathology (Generalizied Anxiety Disorder Scale-7, GAD-7) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 0 to 3 (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day).
  * GAD-7 total score ranges from 0 to 21 (classification of scores: 0 - 4: no to low risk, 5 - 9: mild, 10 - 14: moderate, >= 15 severe).
  * Consequently, a higher score means a worse generalized anxiety disorder psychopathology.
Eating disorder psychopathology (Eating Disorder Examination-Questionnaire-8, EDE-Q-8) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 0 to 6 (0 = characteristic was not present to 6 = characteristic was present every day or in extreme form).
  * Subscale scores (restraint, eating concern, weight concern, shape concern), as well as a total score can be calculated, the total score ranges from 0 to 48.
  * Consequently, a higher score means a worse eating disorder psychopathology.
Social anxiety disorder psychopathology (Mini-Social Phobia Inventory, Mini-SPIN) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 0 to 4 (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = very much, 4 = extremely).
  * Mini-Spin total score ranges from 0 to 12.
  * Consequently, a higher score means a worse social anxiety disorder psychopathology.
Treatment expectation (Generic Rating for Treatment Pre-Experiences, Treatment Expectations, and Treatment Effects, G-EEE) | Baseline, post intervention (after 2 weeks)
  - Items range from 0 to 10 (depending on the item from "no improvement" to "greatest improvement imaginable", from "no worsening" to "greatest worsening imaginable", from "no complaints" to "greatest complaints imaginable") and one item, where previous treatment experience is assessed via a choice of "I have never experienced this treatment." (continue with question 8), "I have experienced this treatment during the last 12 months (nearly) daily.", "I have experienced this treatment during the last 12 months on more than 10 days.", "I have experienced this treatment during the last 12 months on about 5 to 10 days.", I have experienced this treatment during the last 12 months on about 1 to 4 days." And "I have not experienced this treatment during the last 12 months, but I have experienced it before."
Treatment credibility and expectancy (Credibility/Expectancy Questionnaire, CEQ) | Baseline
  * Items range from 1 to 9 (Item 1 of Set 1: 1= not at all logical, 5 = somewhat logical, 9 = very logical, Item 2 of Set 1: 1= not at all useful, 5 = somewhat useful, 9 = very useful, Item 3 of Set 1: 1 = not at all confident, 5 = somewhat confident, 9 = very confident, Item 1 of Set 2: 1 = not at all, 5 = somewhat, 9 = very much), Item 4 of Set 1 and Item 2 of Set 2 give a choice of 0% to 100% in steps of 10 %.
  * CEQ composite score can be derived for each factor (expectancy and credibility)
Trait reward responsiveness (Reward Responsiveness Scale, RRS) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 1 to 4 (1= strong disagreement, 2 = mild disagreement, 3 = mild agreement, 4 = strong agreement)
  * RRS total score ranges from 8 to 32.
  * Consequently, a higher score means a higher reward responsiveness.
Stress level (Perceived-Stress-Scale 10, PSS-10) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 1 to 5 (1= never, 2 = almost never, 3 = sometimes, 4 = fairly often, 5 = very often) Items 4, 5, 7 and 8 are reverse scored for the total score.
  * PH=perceived helplessness subscale; PSE=perceived self-efficacy subscale
  * PH subscale is computed by summing up Items 1, 2, 3, 6, 9 and 10; the PSE subscale is computed by summing up items 4, 5, 7 and 8
  * PSS-10 total score is the sum of all PH and reversed PSE items
  * Consequently, a higher score means a greater level of stress.
Anhedonia (Snaith-Hamilton-Pleasure-Scale, SHAPS-D) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from "Definitely Agree", "Agree", "Disagree", and "Strongly Disagree". Either of the "Disagree responses" receive a score of 1 and either of the "Agree responses" receive a score of 0.
  * SHAPS-D total score ranges from 0 to 14.
  * Consequently, a higher score means a greater state anhedonia.
Depressive expectations (Depressive Expectations Scale, DES) | Baseline, post intervention (after 2 weeks), 4 months follow up
  * Items range from 1 to 5 (1 = I disagree , 2 = I partially disagree, 3 = neutral, 4 = I partially agree, 5 = I agree).
  * DES total score ranges from 25 to 125
  * Consequently, a higher score means more dysfunctional depressive expectations.
Personality traits (Big Five Inventory 10, BFI-10) | Baseline, post intervention (after 2 weeks), up to four months follow up
  * Items range from 1 (disagree strongly) to 5 (agree strongly).
  * Scales: openness to experience, conscientiousness, extraversion, agreeableness and neuroticism

OTHER OUTCOMES:
Adherence | post intervention (after 2 weeks), 4 months follow up
  * Number of completed online surveys regarding the intervention exercises (T1 to T14: daily online surveys over the course of two weeks)
  * Self report of implementation of daily excercises in post intervention survey and follow up survey.
Influence of type of positive activity/type of pleasant situation | during daily excercises (14 days)
  - Type of activities and reflected pleasant situations that have been selected in the daily online surveys (e.g. social, sports ...)
Problems and obstacles during the intervention | post intervention (after 2 weeks), 4 months follow up
  - Frequency of telephone contacts made with the principal contact person (Laura Potsch) and specified problems with the implementation of the daily excercises in the daily online survey
Sociodemographic variables | baseline
  - Gender, age, education, employment, medication, self report lifetime diagnosis of psychiatric conditions, previous experience with psychotherapy etc.
Perceived system usability (System usability Scale, SUS), general feedback about the online intervention | post intervention (after 2 weeks)
  * Items of the SUS range from 1 to 5 (1= strongly disagree to 5 = strongly agree).
  * After a computation, the SUS score can range from 0 to 100. A SUS score above a 68 is considered above average.
  * general feedback about the online intervention: free text entries about the online intervention: criticism, change requests, praise, one closed question: "Would you recommend the online intervention to someone else?" Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Dept. of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Germany
Locations (1):
- Philipps University, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alloy LB, Olino T, Freed RD, Nusslock R. Role of Reward Sensitivity and Processing in Major Depressive and Bipolar Spectrum Disorders. Behav Ther. 2016 Sep;47(5):600-621. doi: 10.1016/j.beth.2016.02.014. Epub 2016 Mar 7. PMID 27816074
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour HJ. Treatment for Anhedonia: A Neuroscience Driven Approach. Depress Anxiety. 2016 Oct;33(10):927-938. doi: 10.1002/da.22490. PMID 27699943
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour H, Rosenfield D. Positive affect treatment for depression and anxiety: A randomized clinical trial for a core feature of anhedonia. J Consult Clin Psychol. 2019 May;87(5):457-471. doi: 10.1037/ccp0000396. PMID 30998048
- [Background] Eshel N, Roiser JP. Reward and punishment processing in depression. Biol Psychiatry. 2010 Jul 15;68(2):118-24. doi: 10.1016/j.biopsych.2010.01.027. Epub 2010 Mar 29. PMID 20303067
- [Background] Geschwind N, Peeters F, Drukker M, van Os J, Wichers M. Mindfulness training increases momentary positive emotions and reward experience in adults vulnerable to depression: a randomized controlled trial. J Consult Clin Psychol. 2011 Oct;79(5):618-28. doi: 10.1037/a0024595. PMID 21767001
- [Background] Kryza-Lacombe M, Pearson N, Lyubomirsky S, Stein MB, Wiggins JL, Taylor CT. Changes in neural reward processing following Amplification of Positivity treatment for depression and anxiety: Preliminary findings from a randomized waitlist controlled trial. Behav Res Ther. 2021 Jul;142:103860. doi: 10.1016/j.brat.2021.103860. Epub 2021 Apr 15. PMID 33894554
- [Background] Linke J, Wessa M. Mental Imagery Training Increases Wanting of Rewards and Reward Sensitivity and Reduces Depressive Symptoms. Behav Ther. 2017 Sep;48(5):695-706. doi: 10.1016/j.beth.2017.04.002. Epub 2017 Apr 18. PMID 28711118
- [Background] Renner F, Ji JL, Pictet A, Holmes EA, Blackwell SE. Effects of Engaging in Repeated Mental Imagery of Future Positive Events on Behavioural Activation in Individuals with Major Depressive Disorder. Cognit Ther Res. 2017;41(3):369-380. doi: 10.1007/s10608-016-9776-y. Epub 2016 Apr 9. PMID 28515538
- [Derived] Potsch L, Rief W. Effectiveness of behavioral activation and mindfulness in increasing reward sensitivity and reducing depressive symptoms - A randomized controlled trial. Behav Res Ther. 2024 Feb;173:104455. doi: 10.1016/j.brat.2023.104455. Epub 2023 Dec 13. PMID 38128402